CLINICAL TRIAL: NCT04988295
Title: A Phase 3, Open-Label, Randomized Study of Amivantamab and Lazertinib in Combination With Platinum-Based Chemotherapy Compared With Platinum-Based Chemotherapy in Patients With EGFR-Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer After Osimertinib Failure
Brief Title: A Study of Amivantamab and Lazertinib in Combination With Platinum-Based Chemotherapy Compared With Platinum-Based Chemotherapy in Patients With Epidermal Growth Factor Receptor (EGFR)-Mutated Locally Advanced or Metastatic Non- Small Cell Lung Cancer After Osimertinib Failure
Acronym: MARIPOSA-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109061; 61186372NSC3002 (Other: Janssen Research & Development, LLC); 2021-001825-33 (EudraCT Number); 2023-506518-33-00 (Registry Identifier: EUCT number)
Expanded Access: NCT04599712 (Approved for marketing)
Record Dates: First submitted 2021-07-30; First posted 2021-08-03 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib; amivantamab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: LACP/ACP-L (Experimental): LACP dosing (study start until 6 November 2022): Participants will receive Lazertinib orally along with Amivantamab, Pemetrexed, and Carboplatin as IV infusion starting on Cycle 1 Day 1 for 4 cycles (each cycle consists of 21 days). After 4 cycles, participants will receive Amivantamab, Pemetrexed and Lazertinib as maintenance until disease progression. ACP-L dosing (from 7 November 2022 until study completion): Participants will receive Amivantamab, Pemetrexed, and Carboplatin starting on Cycle 1 Day 1 for 4 cycles. Lazertinib in ACP-L will start on Cycle 5 Day 1 or sooner if carboplatin is discontinued before cycle 4 (each cycle consists of 21 days). Beginning with Cycle 5 Day 1, participants will receive Amivantamab, Pemetrexed and Lazertinib as maintenance until disease progression.
  Interventions: Drug: Lazertinib; Drug: Amivantamab; Drug: Pemetrexed; Drug: Carboplatin
- Arm B: CP (Carboplatin and Pemetrexed) (Active Comparator): Participants will receive Pemetrexed in combination with Carboplatin as IV infusion for up to 4 cycles (each cycle consists of 21 days). After 4 cycles, participants will receive Pemetrexed as maintenance until disease progression.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin
- Arm C: ACP (Amivantamab, Carboplatin and Pemetrexed) (Experimental): Participants will receive Amivantamab, Pemetrexed, and Carboplatin as IV infusion for up to 4 cycles (each cycle consists of 21 days). After 4 cycles, participants will receive Amivantamab and Pemetrexed as maintenance until disease progression.
  Interventions: Drug: Amivantamab; Drug: Pemetrexed; Drug: Carboplatin
- Arm A2 (Extension Cohort): ACP-L (Experimental): Participants will receive Amivantamab, Pemetrexed and Carboplatin as IV infusion for up to 4 cycles (each cycle consists of 21 days), Lazertinib will start on C5D1 or sooner if carboplatin is discontinued earlier). After 4 cycles, participants will receive Pemetrexed, Amivantamab, Lazertinib as maintenance until disease progression.
  Interventions: Drug: Lazertinib; Drug: Amivantamab; Drug: Pemetrexed; Drug: Carboplatin
- Arm C2 (Extension Cohort): ACP (Experimental): Participants will receive Amivantamab, Pemetrexed, and Carboplatin as IV infusion for up to 4 cycles (each cycle consists of 21 days). After 4 cycles, participants will receive Amivantamab and Pemetrexed as maintenance until disease progression.
  Interventions: Drug: Amivantamab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Lazertinib — Lazertinib will be administered orally.
  Other Names: JNJ-73841937; YH-25448
  Arms: Arm A2 (Extension Cohort): ACP-L; Arm A: LACP/ACP-L
Drug: Amivantamab — Amivantamab will be administered as an IV infusion.
  Other Names: JNJ-61186372
  Arms: Arm A2 (Extension Cohort): ACP-L; Arm A: LACP/ACP-L; Arm C2 (Extension Cohort): ACP; Arm C: ACP (Amivantamab, Carboplatin and Pemetrexed)
Drug: Pemetrexed — Pemetrexed will be administered as an IV infusion.
Drug: Carboplatin — Carboplatin will be administered as an IV infusion.

SUMMARY:
The purpose of this study is to assess the efficacy of adding lazertinib to amivantamab, carboplatin, and pemetrexed (LACP/ACP-L dosing strategies) and amivantamab, carboplatin and pemetrexed (ACP) compared with carboplatin and pemetrexed (CP) in participants with locally advanced or metastatic epidermal growth factor receptor (EGFR) Exon 19del or Exon 21 L858R substitution non-small cell lung cancer (NSCLC) after osimertinib failure. The purpose of the extension cohort is to further describe the safety and efficacy for the ACP-L dosing schedule versus ACP with additional data. After completion of the primary analysis, the study may eventually transition to an open-label extension (OLE) or long-term extension (LTE) phase during which participants will have the option to continue their assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have at least 1 measurable lesion, according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, that has not been previously irradiated
* Participant must have histologically or cytologically confirmed, locally advanced or metastatic, non-squamous non-small cell lung cancer (NSCLC), characterized at or after the time of locally advanced or metastatic disease diagnosis by either epidermal growth factor receptor (EGFR) Exon 19del or Exon 21 L858R mutation
* A participant with a history of brain metastases must have had all lesions treated as clinically indicated (that is, no current indication for further definitive local therapy). Any definitive local therapy to brain metastases must have been completed at least 14 days prior to randomization and the participant can be receiving no greater than10 milligrams (mg) prednisone or equivalent daily for the treatment of intracranial disease
* Participant must have Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Any toxicities from prior systemic anticancer therapy must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Grade 1 or baseline level (except for alopecia [any grade], Grade <= 2 peripheral neuropathy, or Grade <= 2 hypothyroidism stable on hormone replacement)
* A participant of childbearing potential must have a negative serum pregnancy test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study
* Participant must have progressed on or after osimertinib monotherapy as the most recent line of treatment. Osimertinib must have been administered as either the first-line treatment for locally advanced or metastatic disease or in the second- line setting after prior treatment with first- or second-generation EGFR tyrosine kinase inhibitor (TKI) as a monotherapy. Participants who received either neoadjuvant and/or adjuvant treatment of any type are eligible if progression to locally advanced or metastatic disease occurred at least 12 months after the last dose of such therapy and then the participant progressed on or after osimertinib in the locally advanced or metastatic setting. Treatment with osimertinib must be discontinued at least 8 days (4 half-lives) prior to randomization (that is last dose no later than Day -8)

Exclusion Criteria:

* Participant received radiotherapy for palliative treatment of NSCLC less than 14 days prior to randomization
* Participant with symptomatic or progressive brain metastases
* Participant has history of or current evidence of leptomeningeal disease, or participant has spinal cord compression not definitively treated with surgery or radiation
* Participant has known small cell transformation
* Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis
* Participant has a history of clinically significant cardiovascular disease including, but not limited to diagnosis of deep vein thrombosis or pulmonary embolism within 4 weeks prior to randomization; myocardial infarction; unstable angina; stroke; transient ischemic attack; coronary/peripheral artery bypass graft; or acute coronary syndrome. Participant has a significant genetic predisposition to venous thromboembolic events. Participant has a prior history of venous thromboembolic events and is not on appropriate therapeutic anticoagulation as per National Comprehensive Cancer Network or local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (247):
- United States (28):
  - Southern Cancer Center, PC, Mobile, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - City of Hope, Duarte, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - TriHealth Network, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - Texas Oncology, Grapevine, Texas
  - Oncology Consultants Texas, Houston, Texas
  - Texas Oncology - Northeast, Longview, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Cancer Care, Wytheville, Virginia
  - NorthWest Medical Specialties, PLLC, Puyallup, Washington
  - Compass Oncology, Vancouver, Washington
- Argentina (8):
  - CINME Centro de Investigaciones Metabolicas, Caba
  - IADT Instituto Argentino de Diagnostico y Tratamiento, CABA
  - Centro Medico Fleischer, CABA
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), CABA
  - Cemaic Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Hospital Privado Universitario De Cordoba, Córdoba
  - Hospital Privado de la Comunidad, Mar del Plata
  - Clínica Viedma, Viedma
- Belgium (7):
  - Grand Hopital De Charleroi Site Les Viviers, Charleroi
  - UZA, Edegem
  - UZ Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - UZ Leuven, Leuven
  - CHU Sart-Tilman, Liège
  - Clinique Saint Pierre, Ottignies
- Brazil (21):
  - Cetus Oncologia, Belo Horizonte
  - CIONC Centro Integrado de Oncologia de Curitiba, Curitiba
  - Ynova Pesquisa Clinica, Florianópolis
  - Fundacao Sao Francisco Xavier, Ipatinga
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Hospital Sao Rafael, Salvador
  - CEPHO Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Hospital Paulistano, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Hospital Nove de Julho, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Onco Star SP Oncologia Ltda, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - COT - Centro Oncologico do Triangulo S.A, Uberlândia
- Bulgaria (4):
  - Multifunctional Hospital for Active Treatment 'Serdika', Sofia
  - Multiprofile Hospital for Active Treatment 'Tokuda Hospital Sofia', Sofia
  - Specialized Hospital for Active Treatment in Oncology, Sofia
  - UMHAT Sofia Med, Sofia
- Canada (3):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - McGill University Health Centre, Montreal, Quebec
- China (31):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chest hospital, Capital medical university, Beijing
  - Hunan Cancer hospital, Changsha
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Southwest Hospital, Chongqing
  - Daping Hospital Army Characteristic Medical Center, Chongqing
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Sun Yat-Sen Memorial Hospital Sun Yat-sen University, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Municipal Central Hospital, Huizhou
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Affiliated Hospital of North Sichuan Medical College, Nanchong
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shenzhen university General Hospital, Shenzhen
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- Czechia (3):
  - Fakultni nemocnice Olomouc - I.P.Pavlova 6, Olomouc
  - Vitkovicka nemocnice a.s., Ostrava- Vitkovice
  - Fakultni nemocnice Plzen, Pilsen
- Rigshospitalet, Copenhagen, Denmark
- France (13):
  - Institut Sainte Catherine, Avignon
  - Hospices Civils de Lyon HCL, Bron
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - Centre Hospitalier du Mans, Le Mans
  - CHR Hôpital Calmette, Lille
  - Hopital Nord, Marseille
  - CHU de Montpellier - Arnaud de Villeneuve, Montpellier
  - Institut Curie, Paris
  - CHU Bordeaux, Pessac
  - CHRU Hopital de Pontchaillou, Rennes
  - CHU Nantes, Sain-Herblain
  - Nouvel Hopital Civil - CHU Strasbourg, Strasbourg
  - CHU Bretonneau, Tours
- Germany (9):
  - Evangelische Lungenklinik Berlin, Berlin
  - Asklepios Klinikum Harburg, Hamburg
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Onkologische Schwerpunktpraxis, Heilbronn
  - POIS Sachsen GmbH iG, Leipzig
  - Bethanien Krankenhaus, Moers
  - Klinikum der Universitaet Muenchen, München
  - Oncologianova GmbH, Recklinghausen
  - Universitaetsklinikum Regensburg, Regensburg
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (8):
  - Health Care Global Enterprises pvt Ltd, Bangalore
  - Artemis Hospital, Gurugram
  - Tata Medical Center, Kolkata
  - Tata Memorial Hospital, Mumbai
  - HCG Manavta Cancer Centre, Nashik
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delh
  - Noble Hospital Pvt Ltd, Pune
  - Bhaktivedanta Hospital & Research Institute, Thane
- Israel (7):
  - Soroka University Medical Center, Beersheba
  - Rambam Health Corporation, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - CRO IRCCS Istituto Nazionale Tumori, Aviano
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero-Universitaria Di Parma, Parma
  - Ospedale S. Maria Delle Croci, Ravenna
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Policlinico G.B.Rossi, Verona
- Japan (15):
  - National Hospital Organization Shibukawa Medical Center, Gunma
  - Hyogo Cancer Center, Hyōgo
  - Kanagawa Cancer Center, Kanagawa
  - Kobe City Medical Center General Hospital, Kobe
  - Kurume University Hospital, Kurume
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Ehime University Hospital, Toon-shi
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Iwakuni Clinical Center, Yamaguchi
  - National Hospital Organization Yamaguchi Ube Medical Center, Yamaguchi
- Malaysia (5):
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Beacon Hospital Sdn Bhd, Petaling Jaya
  - Subang Jaya Medical Centre, Subang Jaya
  - Mount Miriam Cancer Hospital, Tanjung Bungah
- Mexico (5):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - CIMOVA, Morals Vargas Centro de Investigación SC, León
  - Health Pharma Professional Research, México
  - Instituto Nacional de Cancerologia, México
  - Oncologia Integral Satelite, Naucalpan
- Netherlands (3):
  - VUMC Amsterdam, Amsterdam
  - Ziekenhuis St Jansdal, Harderwijk
  - Erasmus MC, Rotterdam
- Poland (7):
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandow, Poznan
  - Private Specialist Hospitals - MedPolonia, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (4):
  - Uls Santa Maria - Hosp. Pulido Valente, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Uls Santo Antonio - Hosp. Santo Antonio, Porto
  - Instituto Portugues de Oncologia, Porto
- Pan American Center for Oncology Trials LLC, Rio Piedras, Puerto Rico
- Russia (2):
  - City Clinical Hospital #1, Nal'chik
  - Llc, Eurocityclinic, Saint Petersburg
- South Korea (9):
  - National Cancer Center, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - GyeongSang National University Hospital, Gyeongsangnam-do
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (17):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp Regional Univ de Malaga, Málaga
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Gral. Univ. Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Linkoping University Hospital, Linköping
  - Skanes universitetssjukhus, Lund
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (10):
  - Adana City Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakirkoy Training and Research Hospital, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Medical Point, Izmir
- United Kingdom (6):
  - Velindre Hospital, Cardiff
  - Edinburgh Cancer Centre Western General, Edinburgh
  - UCL Cancer Institute, London
  - Guys and St Thomas NHS Foundation Trust, London
  - The Royal Marsden NHS Trust, London
  - The Christie Nhs Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 657 participants were enrolled in the main study. During the study, a separate open-label randomized extension cohort was added. A total of 119 participants were enrolled into the extension cohort. Main study results are alone reported for primary completion date (PCD; 10-July-2023).
Pre-assignment Details: At the time of PCD, extension cohort enrollment was still ongoing. As per protocol, extension cohort analysis was not included as part of main study primary analysis. Currently no information other than total count of participants for extension cohort is available and for reporting purpose extension cohort arms (A2 and C2) have been combined in the table. Results of extension cohort will be reported later, upon completion of analysis, at which point arms A2 and C2 details will be reported.
Groups:
- Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L): Schedule 1:LACP:study start to 06-Nov-2022:Lazertinib 240 milligrams(mg) orally daily along with amivantamab and chemotherapy (carboplatin and pemetrexed). Amivantamab 1400 mg (1750 mg if body weight>= 80 kilograms[kg]) intravenous(IV) infusion on Cycle 1 Days 1/2, 8 and 15 and Cycle 2 Day 1 and then 1750 mg (2100 mg if body weight >=80 kg) on Day 1 of each 21-day cycle, starting at cycle 3. Participants received chemotherapy:pemetrexed 500 milligrams per meter square(mg/m^2) IV infusion on Day 1 of each 21-day cycle, along with carboplatin area under concentration-time curve of 5 (AUC 5) IV infusion on Day 1 for up to 4 cycles and then as maintenance monotherapy until disease progression(DP). Schedule 2:ACP-L:07-Nov-2022 to study end:Amivantamab 1400 mg (1750 mg if body weight>=80 kg) IV infusion on Cycle 1 Days 1/2, 8 and 15 and Cycle 2 Day 1 and then 1750 mg (2100 mg if body weight >=80 kg) on Day 1 of each 21-day cycle, starting at cycle 3. Participants also received chemotherapy:pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle, along with carboplatin AUC 5 IV infusion on Day 1 for up to 4 cycles and then as maintenance monotherapy until DP. Lazertinib was administered 240 mg orally, once daily starting Cycle 5 Day 1 or sooner if carboplatin was discontinued earlier. In both schedules, Lazertinib, amivantamab and pemetrexed:continued until DP, participant withdrawal, adverse event, investigator's decision/initiation of new systemic anti-cancer treatment.
- Main Study: Arm B: Carboplatin + Pemetrexed (CP): Participants received chemotherapy with pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle, in combination with carboplatin area under the concentration-time curve of 5 mg/mL per minute (AUC 5) was administered as an IV infusion on Day 1, for up to 4 cycles, and then as maintenance monotherapy until disease progression, participant consent withdrawal, adverse event, investigator's decision, or initiation of new systemic anti-cancer treatment.
- Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP): Participants received amivantamab 1400 mg (1750 mg if body weight is >= 80 kg) by IV infusion once weekly starting from Cycle 1 Days 1/2, 8, and 15, and Cycle 2 Day 1, then 1750 mg (2100 mg if body weight is >=80 kg) on Day 1 of each 21-day cycle, starting with Cycle 3. Participants also received chemotherapy with pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle, in combination with carboplatin area under the concentration-time curve of 5 mg/mL per minute (AUC 5) was administered as an IV infusion on Day 1, for up to 4 cycles. Amivantamab and pemetrexed treatments were to be continued until disease progression, participant consent withdrawal, adverse event, investigator's decision, or initiation of new systemic anti-cancer treatment.
- Extension Cohort: All Participants (Arm A2 [ACP-L] + C2 [ACP]): In Arm A2, participants received amivantamab 1400 mg (1750 mg if body weight>=80 kg) IV infusion once weekly from Cycle 1 Days 1/2, 8, and 15, and Cycle 2 Day 1, and then 1750 mg (2100 mg if body weight >=80 kg) on Day 1 of each 21-day cycle, starting at cycle 3. Participants also received chemotherapy: pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle, in combination with carboplatin area under concentration-time curve of 5 mg/mL per minute (AUC 5) IV infusion administered on Day 1 for up to 4 cycles. Lazertinib was administered 240 mg orally, once daily starting Cycle 5 Day 1 or sooner if carboplatin was discontinued earlier. Amivantamab, pemetrexed and lazertinib were to be continued until disease progression (DP), participant withdrawal, adverse event (AE), investigator's decision or initiation of new systemic anti-cancer treatment. In Arm C2, participants received amivantamab 1400 mg (1750 mg if body weight >=80 kg) IV infusion once weekly from Cycle 1 Days 1/2, 8, and 15, and Cycle 2 Day 1, then 1750 mg (2100 mg if body weight is >=80 kg) on Day 1 of each 21-day cycle, starting with Cycle 3. Participants also received chemotherapy: pemetrexed 500 mg/m^2 IV infusion on Day 1 of each 21-day cycle, in combination with carboplatin AUC 5 IV infusion was administered on Day 1, for up to 4 cycles. Amivantamab and pemetrexed were to be continued until DP, participant withdrawal, AE, investigator's decision or initiation of new systemic anti-cancer treatment.
Period: Overall Study
Arm/Group | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP) | Extension Cohort: All Participants (Arm A2 [ACP-L] + C2 [ACP])
Started | 263 | 263 | 131 | 119
Treated (Safety Analysis Set) | 263 | 243 | 130 | 119
Completed (As per protocol, participants who died were also considered as completed) | 67 | 65 | 26 | 0
Not Completed | 196 | 198 | 105 | 119
Not completed — Withdrawal by Subject | 9 | 29 | 6 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Study participation ongoing | 186 | 169 | 99 | 119

BASELINE CHARACTERISTICS:
Population: Only main study (N=657) results are reported, thus column "Total participants" presents main study data. Per protocol, extension cohort analysis was not included in main study primary analysis. Extension cohort results will be reported later, upon analysis completion, at which point arms A2 and C2 details will be reported. For reporting purpose of extension cohort at this time since data is still not available, single combined arm for extension cohort (A2/C2) is presented with '0' participants.
Groups:
- Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L): LACP dosing (study start until 6 November 2022): Participants received Lazertinib 240 milligrams (mg) orally on Day 1 of each subsequent cycle, starting with Cycle 3, along with Amivantamab 1400 mg (1750 mg if body weight greater than or equal to [>=80] kilograms [kg]) on Cycle 1 Days 1, 2, 8, and 15, and Cycle 2 Day 1 and 1750 mg (2100 mg if body weight >=80 kg). Participant also received Pemetrexed 500 mg per square meter (mg/m^2) on Day 1 21-day cycle, in combination with carboplatin 750 mg as IV infusion starting on Cycle 1 Day 1 for 4 cycles. From cycle 5 onwards, participants received Amivantamab, Pemetrexed and Lazertinib IV infusions at same dose, as maintenance until disease progression. ACP-L dosing (from 7 November 2022 until study completion): Participants received Amivantamab 1400 mg (1750 mg if body weight >=80] kg) on Cycle 1 Days 1,2, 8, and 15, and Cycle 2 Day 1 and 1750 mg (2100 mg if body weight >=80 kg). Participant also received Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle, in combination with carboplatin 750 mg as IV infusion starting on Cycle 1 Day 1 for 4 cycles. Lazertinib 240 mg in ACP-L started on Cycle 5 Day 1 or sooner if carboplatin is discontinued before cycle 4. From cycle 5 onwards, participants received Amivantamab, Pemetrexed and Lazertinib IV infusions at same dose, as maintenance until disease progression. Each cycle consists of 21 days.
- Main Study: Arm B: Carboplatin + Pemetrexed (CP): Participants received Pemetrexed 500 mg/m^2 IV infusion and carboplatin 750 mg IV infusion from Day 1 of Cycle 1 to 4. From cycle 5 onwards, participants received Pemetrexed 500 mg/m^2 IV infusion, as maintenance until disease progression. Each cycle consists of 21 days.
- Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP): Participants received Amivantamab 1400 mg (1750 mg if body weight >=80 kg) on Cycle 1 Days 1,2, 8, and 15, and Cycle 2 Day 1 and 1750 mg (2100 mg if body weight >=80 kg) on Day 1 of each cycle, starting with Cycle 3. Participants also received Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle, in combination with carboplatin 750 mg as IV infusion starting on Cycle 1 Day 1 for 4 cycles. From cycle 5 onwards, participants received Amivantamab and Pemetrexed IV infusions at same dose, as maintenance until disease progression. Each cycle consists of 21 days.
- Total: Total of all reporting groups
Arm/Group | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP) | Extension Cohort: All Participants (Arm A2 [ACP-L] + C2 [ACP]) | Total
Number analyzed (Participants) | 263 | 263 | 131 | 0 | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.96) | 60.6 (10.13) | 61.2 (10.06) |  | 60.6 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 157 | 81 |  | 406
  Male | 95 | 106 | 50 |  | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 9 |  | 54
  Not Hispanic or Latino | 234 | 234 | 118 |  | 586
  Unknown or Not Reported | 7 | 6 | 4 |  | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 |  | 4
  Asian | 125 | 127 | 63 |  | 315
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 4 | 1 | 3 |  | 8
  White | 129 | 123 | 60 |  | 312
  More than one race | 0 | 2 | 0 |  | 2
  Unknown or Not Reported | 5 | 7 | 4 |  | 16
Region of Enrollment [Count of Participants; unit: Participants] — Population: For extension cohort, data was not available at the time of primary analysis results reporting. Hence, enrollment data was reported only for main study.
  Participants
    ARGENTINA | 5 | 6 | 0 |  | 11
    BELGIUM | 10 | 3 | 3 |  | 16
    BRAZIL | 10 | 13 | 6 |  | 29
    BULGARIA | 0 | 1 | 1 |  | 2
    CANADA | 7 | 11 | 4 |  | 22
    CHINA | 45 | 40 | 15 |  | 100
    CZECH REPUBLIC | 1 | 1 | 1 |  | 3
    FRANCE | 14 | 18 | 7 |  | 39
    GERMANY | 3 | 4 | 0 |  | 7
    HONG KONG | 0 | 2 | 0 |  | 2
    INDIA | 14 | 8 | 4 |  | 26
    ISRAEL | 6 | 4 | 3 |  | 13
    ITALY | 20 | 19 | 11 |  | 50
    JAPAN | 17 | 24 | 9 |  | 50
    MALAYSIA | 4 | 5 | 8 |  | 17
    MEXICO | 5 | 4 | 2 |  | 11
    NETHERLANDS | 1 | 4 | 2 |  | 7
    POLAND | 1 | 9 | 4 |  | 14
    PORTUGAL | 4 | 2 | 1 |  | 7
    RUSSIAN FEDERATION | 1 | 0 | 0 |  | 1
    SOUTH KOREA | 25 | 21 | 17 |  | 63
    SPAIN | 30 | 24 | 13 |  | 67
    SWEDEN | 3 | 1 | 0 |  | 4
    TAIWAN | 10 | 17 | 7 |  | 34
    TURKEY | 10 | 5 | 4 |  | 19
    UNITED KINGDOM | 8 | 10 | 2 |  | 20
    UNITED STATES | 9 | 7 | 7 |  | 23

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization until the date of objective disease progression or death, whichever came first, as assessed by BICR according to RECIST version 1.1. Progressed disease: Sum of diameters increased by greater than or equal to (>=)20 percent (%) and >=5 millimeter (mm) from nadir (including baseline if it was smallest sum).
Time Frame: From randomization to either disease progression or death, whichever occurred first (up to 1 year 7 months)
Population: Full analysis set (FAS) as defined in the protocol included all randomized participants, classified according to their assigned treatment arm regardless of the actual treatment received. The outcomes reported here are for main study participants. For Arm A participants, data were planned to be analyzed as a single arm collectively for the LACP and ACP-L dosing regimens.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP)
Number analyzed (Participants) | 263 | 263 | 131
months | 8.31 [6.77 to 9.10] | 4.17 [4.04 to 4.44] | 6.28 [5.55 to 8.41]
Statistical Analysis 1: Comparison: Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) vs Main Study: Arm B: Carboplatin + Pemetrexed (CP); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.35 to 0.56]
Statistical Analysis 2: Comparison: Main Study: Arm B: Carboplatin + Pemetrexed (CP) vs Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.48, 95% CI [0.36 to 0.64]

2. Primary Outcome: Main Study + Extension Cohort: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Follow-up for the extension cohort is still ongoing and thus results from the analysis that includes the extension cohort will be reported up on study completion.
Time Frame: up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

3. Secondary Outcome: Main Study+ Extension Cohort: Objective Response Rate as Assessed by Blinded Independent Central Review
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

4. Secondary Outcome: Main Study+ Extension Cohort: Overall Survival
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

5. Secondary Outcome: Main Study+ Extension Cohort: Duration of Response as Assessed by Blinded Independent Central Review
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

6. Secondary Outcome: Main Study+ Extension Cohort: Time to Subsequent Therapy
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

7. Secondary Outcome: Main Study+ Extension Cohort: Progression-free Survival (PFS) After First Subsequent Therapy (PFS2)
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

8. Secondary Outcome: Main Study+ Extension Cohort: Time to Symptomatic Progression
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

9. Secondary Outcome: Main Study+ Extension Cohort: Intracranial Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

10. Secondary Outcome: Main Study: Number of Participants With Adverse Events (AEs)
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

11. Secondary Outcome: Main Study+ Extension Cohort: Number of Participants With Adverse Events (AEs) by Severity
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

12. Secondary Outcome: Main Study+ Extension Cohort: Number of Participants With Clinical Laboratory Abnormalities
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

13. Secondary Outcome: Main Study+ Extension Cohort: Serum Concentration of Amivantamab
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

14. Secondary Outcome: Main Study+ Extension Cohort: Plasma Concentration of Lazertinib
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

15. Secondary Outcome: Main Study + Extension Cohort: Number of Participants With Serum Anti-amivantamab Antibodies
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

16. Secondary Outcome: Main Study+ Extension Cohort: Change From Baseline With Non-Small Cell Lung Cancer - Symptom Assessment Questionnaire (NSCLC-SAQ)
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

17. Secondary Outcome: Main Study+ Extension Cohort: Change From Baseline With European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

18. Secondary Outcome: Main Study+ Extension Cohort: Change From Baseline With Patient-Reported Outcomes Measurement Information System -Physical Function (PROMIS-PF)
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

19. Primary Outcome: Main Study + Extension Cohort: Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review
Time Frame: Up to 4 years 10 months
Reporting Status: Not Posted, anticipated posting 2027-09

ADVERSE EVENTS:
Time Frame: From Cycle 1 Day 1 up to 1 year 7 months
Description: SAEs & Other AEs:safety set-randomized participants who had at least 1 dose of study drug. All-cause mortality:FAS-all randomized participants, classified per assigned drug regardless of actual drug received. As per statistical analysis, Arm A AE planned to be collected and analyzed as single arm regardless of regimen LACP/ACP-L received. Since extension cohort is ongoing and its data collection and analysis was not planned for primary analysis, AE data will be reported after study completion.
Arm/Group | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP)
All-Cause Mortality (participants affected / at risk) | 69/263 | 65/263 | 27/131
Serious Adverse Events (participants affected / at risk) | 137/263 | 49/243 | 42/130
Other Adverse Events (participants affected / at risk) | 261/263 | 222/243 | 129/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) (N=263) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) (N=243) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP) (N=130)
Sepsis (Infections and infestations) | 6 | 1 | 3
Covid-19 (Infections and infestations) | 6 | 0 | 2
Skin Infection (Infections and infestations) | 1 | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 1
Infectious Pleural Effusion (Infections and infestations) | 0 | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 2 | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Coronavirus Pneumonia (Infections and infestations) | 1 | 0 | 0
Covid-19 Pneumonia (Infections and infestations) | 1 | 0 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 3 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 5 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0
Septic Shock (Infections and infestations) | 2 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 5 | 4
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 20 | 5 | 2
Myelosuppression (Blood and lymphatic system disorders) | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 21 | 6 | 2
Leukopenia (Blood and lymphatic system disorders) | 10 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 1
Nausea (Gastrointestinal disorders) | 8 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 3 | 2
Fatigue (General disorders) | 1 | 1 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 2 | 0
General Physical Health Deterioration (General disorders) | 1 | 0 | 0
Localised Oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 3 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Sudden Death (General disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 2
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 9 | 0 | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 4 | 1 | 2
Embolism (Vascular disorders) | 4 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic Cytolysis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 3 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 0
General Physical Condition Abnormal (Investigations) | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0 | 0
Troponin I Increased (Investigations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 1 | 1
Optic Neuritis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0
Subdural Hygroma (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
Bladder Dilatation (Renal and urinary disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 1
Aseptic Pustule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Arm A: Lazertinib + Amivantamab + Carboplatin + Pemetrexed (LACP/ACP-L) (N=263) | Main Study: Arm B: Carboplatin + Pemetrexed (CP) (N=243) | Main Study: Arm C: Amivantamab + Carboplatin + Pemetrexed (ACP) (N=130)
Nausea (Gastrointestinal disorders) | 130 | 90 | 58
Constipation (Gastrointestinal disorders) | 96 | 72 | 50
Stomatitis (Gastrointestinal disorders) | 120 | 21 | 41
Vomiting (Gastrointestinal disorders) | 75 | 42 | 31
Diarrhoea (Gastrointestinal disorders) | 66 | 16 | 17
Abdominal Pain (Gastrointestinal disorders) | 13 | 6 | 7
Dry Mouth (Gastrointestinal disorders) | 6 | 1 | 7
Haemorrhoids (Gastrointestinal disorders) | 22 | 1 | 7
Neutropenia (Blood and lymphatic system disorders) | 173 | 98 | 73
Thrombocytopenia (Blood and lymphatic system disorders) | 156 | 69 | 57
Anaemia (Blood and lymphatic system disorders) | 141 | 96 | 50
Leukopenia (Blood and lymphatic system disorders) | 106 | 67 | 37
Lymphopenia (Blood and lymphatic system disorders) | 36 | 20 | 12
Rash (Skin and subcutaneous tissue disorders) | 125 | 12 | 56
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 62 | 7 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 17 | 20
Dry Skin (Skin and subcutaneous tissue disorders) | 22 | 4 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 8 | 8
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 16 | 4 | 3
Skin Ulcer (Skin and subcutaneous tissue disorders) | 15 | 0 | 1
Oedema Peripheral (General disorders) | 85 | 15 | 42
Fatigue (General disorders) | 69 | 47 | 35
Asthenia (General disorders) | 67 | 39 | 34
Pyrexia (General disorders) | 29 | 24 | 13
Malaise (General disorders) | 17 | 10 | 5
Infusion Related Reaction (Injury, poisoning and procedural complications) | 142 | 1 | 74
Decreased Appetite (Metabolism and nutrition disorders) | 85 | 50 | 40
Hypoalbuminaemia (Metabolism and nutrition disorders) | 104 | 21 | 29
Hypokalaemia (Metabolism and nutrition disorders) | 54 | 15 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 23 | 10 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 44 | 9 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 33 | 9 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 40 | 16 | 13
Paronychia (Infections and infestations) | 132 | 1 | 48
Covid-19 (Infections and infestations) | 39 | 25 | 25
Conjunctivitis (Infections and infestations) | 11 | 5 | 10
Folliculitis (Infections and infestations) | 9 | 0 | 8
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 4 | 8
Urinary Tract Infection (Infections and infestations) | 22 | 6 | 3
Alanine Aminotransferase Increased (Investigations) | 55 | 67 | 26
Aspartate Aminotransferase Increased (Investigations) | 43 | 57 | 19
Weight Decreased (Investigations) | 31 | 17 | 14
Blood Alkaline Phosphatase Increased (Investigations) | 24 | 13 | 9
Gamma-Glutamyltransferase Increased (Investigations) | 26 | 25 | 7
Blood Creatinine Increased (Investigations) | 31 | 14 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 29 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 17 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 35 | 7 | 11
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 28 | 6 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 23 | 18 | 13
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 11 | 7 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 9 | 8
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 7
Headache (Nervous system disorders) | 23 | 28 | 11
Dizziness (Nervous system disorders) | 32 | 15 | 10
Peripheral Sensory Neuropathy (Nervous system disorders) | 22 | 6 | 5
Dysgeusia (Nervous system disorders) | 17 | 8 | 4
Paraesthesia (Nervous system disorders) | 19 | 6 | 3
Deep Vein Thrombosis (Vascular disorders) | 19 | 3 | 8
Hypotension (Vascular disorders) | 16 | 5 | 3
Insomnia (Psychiatric disorders) | 15 | 7 | 10
Dry Eye (Eye disorders) | 12 | 2 | 7
Hyperbilirubinaemia (Hepatobiliary disorders) | 18 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study site and investigator shall not publish study results except as required by law or as specified in a separate, written agreement between the sponsor and the study site or the investigator.

DOCUMENTS (2):
  • Study Protocol (2024-04-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT04988295/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT04988295/SAP_001.pdf